CLINICAL TRIAL: NCT04676490
Title: Recordable Cards for Optimizing Outcomes and Reducing Disparities After ED Discharge
Brief Title: The RECORD-ED Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, K. Casey Lion, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00002727
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Asthma in Children

STUDY DESIGN:
Intervention Model Description: This is behavioral intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Discharge Care (No Intervention): Usual ED discharge care
- RECORD-ED Card (Experimental): Usual care, plus a physical greeting card-style card with audio discharge instructions (English or Spanish) recorded on it
  Interventions: Other: RECORD-ED Card
- RECORD-ED Patient Portal (Experimental): Usual care, plus access to audio-recorded discharge instructions (English or Spanish) through the patient portal
  Interventions: Other: RECORD-ED Patient Portal

INTERVENTIONS:
Other: RECORD-ED Card — Low-cost and low-tech recordable audio card containing language-concordant discharge instructions for families of children under age 10 presenting to the ED for asthma exacerbations with no or public insurance and a preference for English or Spanish. Recordable cards allow for multiple audio reviews of the instructions by multiple caregivers without dependence on access to the internet or smartphone technologies.
  Arms: RECORD-ED Card
Other: RECORD-ED Patient Portal — Audio recorded, language concordant discharge instructions via patient portal
  Arms: RECORD-ED Patient Portal

SUMMARY:
In this pilot randomized trial, the investigators will evaluate the feasibility, acceptability, and potential family-centered outcomes associated with providing asthma discharge instructions in audio-recorded format in addition to written format, compared to written instructions alone. The study will enroll 100 families of children being discharged home from an emergency department visit, who prefer either English or Spanish for medical care, and assess outcomes at 3 time-points.

DETAILED DESCRIPTION:
This pilot randomized controlled trial seeks to test the feasibility and acceptability of providing and evaluating outcomes associated with audio-recorded, language concordant ED discharge instructions (the RECORD-ED intervention) among low-income parents of children treated for an asthma exacerbation. The study will enroll 100 children and their parent/caregiver with low income and/or limited English proficiency (LEP) who are being discharged home from the emergency department (ED) with a diagnosis of asthma; 20 will be randomized to receive usual discharge care, 40 will receive a physical card with audio-recorded discharge instructions, in addition to usual care, and another 40 will receive access to audio-recorded instructions through the patient portal in addition to usual care. The study team will also send a brief survey to providers and nurses in the ED about the intervention, and conduct qualitative interviews with parents and nurses about their experiences using the recordable cards for discharge instructions. Primary outcomes will focus on feasibility and acceptability of the intervention and outcome ascertainment protocols, as recommended for pilot studies. Parents will complete surveys at 3 time points. Parent outcomes (instruction recall, adherence, comfort with home care, caregiver quality of life), child outcomes (asthma control, including rescue medication use and school absence if age-appropriate), and follow-up utilization (primary care follow-up, 3-month ED and hospital re-visits) will be collected to inform planning for the subsequent R01 proposal.

ELIGIBILITY:
Main pilot RCT: This study will enroll children and their parents who meet the following criteria:

* child age 10 years old or younger
* child with public or no insurance
* child being discharged home from the ED with discharge instructions for asthma/reactive airways disease
* parent with a preferred language for medical care of English or Spanish
* parent/caregiver present in the ED is child's legal guardian
* parent reports access to a telephone (including landline or non-smartphone) for completing follow-up surveys

Parent interviews: Parents will be eligible for the qualitative interviews if they meet the following criteria:

* enrolled in pilot RCT
* randomized to RECORD-ED arm
* completed second follow-up survey within 10 days of ED visit and can complete interview within 14 days of visit
* parent language, literacy (based on single item literacy screener question), and previous experience with ED visits for asthma will be used to purposively sample an even number of English- and Spanish-speaking parents

Provider and nurse surveys: Providers and nurses in the ED will be eligible for the post-visit survey if they meet the following criteria:

-involved in caring for an enrolled patient, randomized to either intervention arm, around the time of discharge

Provider and nurse interviews: Providers and nurses will be eligible for an interview if they meet the following criteria:

-involved in discharge for 1 or more patients in either intervention arm over the past month, with at least one in the past 14 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Protocol feasibility | 3 months after ED visit
  [The protocol will be determined to be feasible if the following criteria are met:
  * successful enrollment of 100 families over 15 months
  * participant retention >70% through 3 follow-up surveys
  * successful ascertainment of parent, child, and utilization outcomes, with <10% of data missing for each outcome (from among those who completed the relevant survey).]

SECONDARY OUTCOMES:
Instruction recall | 2 days after
  Caregiver-reported discharge instructions, in 5 domains (home care, medications [including over-the-counter], expected illness progression, follow-up, and return precautions), will be compared to chart-abstracted instructions and coded for concordance (fully or mostly concordant (3), partially concordant (2), minimally concordant (1), or wrong/ not concordant (0)). Overall instruction recall concordance will be calculated as the percent of domains that were fully or mostly concordant.
Comfort with home care | 2 days after ED visit
  These 8 caregiver-reported care transition items pertain to having received enough information; knowing warning signs; understanding how to manage the child's care; knowing who to call; the child being healthy enough to go home; having an easily understood plan; understanding the purpose of each medication; and understanding how much and how often to give each medication. Responses are on a Likert scale, from "strongly disagree" (1) to "strongly agree" (5)
PCP follow-up | 1 week after ED visit
  Caregivers will be asked to report on any visits to the PCP since the ED visit, and whether the visit was specifically for the condition that prompted the initial ED visit. The response will be coded as yes or no.
Asthma Caregiver Quality of Life | 1 week after ED visit
  We will use the Pediatric Asthma Caregiver's Quality of Life Questionnaire to measure the current impact of the child's asthma symptoms and management on caregiver QoL. This 13-item measure captures asthma-related caregiver stress, uncertainty, sleep disruption and activity limitation; it is associated with child asthma control and life stress, and exhibits good responsiveness to intervention.
Provider-rated intervention acceptability | Within 3 days of ED visit
  We will use the 4-item Acceptability of Intervention measure to capture nurses' and providers' assessment of the acceptability of a recordable card for discharge instructions. Responses are using a 5-point Likert scale. The survey to assess this measure will be brief and anonymous, sent to nurses and providers recorded as having been part of discharge for families randomized to the intervention arm.
Child asthma control | 3 months after ED visit
  Child asthma control will be measured using the Test for Respiratory and Asthma Control in Kids (TRACK, age <=4 years) or the Asthma Therapy Assessment Questionnaire (ATAQ, age 5-10 years) control domain, depending on child age at enrollment. The TRACK includes 5 questions assessing parent-reported symptoms, nighttime awakenings, activity interference, rescue medication use, and oral corticosteroid use. It produces a scale score (0-100), with scores <80 indicating poorly controlled asthma. The ATAQ control domain includes 7 questions, each dichotomously scored and summed, assessing parent-reported symptoms, nighttime awakenings, activity interference, rescue medication use, and missed school. It produces scores 0-7, with higher scores reflecting worse asthma control.
ED and hospital re-visits | 3 months after ED visit
  Number of visits to ED and/or overnight hospital stays since index ED visit; collected via parent-report and from administrative data.
Medication adherence | 2 days after ED visit
  This outcome is coded as correct or incorrect, based on comparing parent-reported actual medication administration (elicited through detailed interview prompts) to EMR-abstracted instructions

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's, Seattle, Washington, United States